CLINICAL TRIAL: NCT03395405
Title: A Phase 2 Multi-Center, Prospective, Randomized, Double-Blind Study to Assess the Clinical and Antiviral Efficacy and Safety of Nitazoxanide for the Treatment of Norovirus in Hematopoietic Stem Cell and Solid Organ Transplant Recipients
Brief Title: NNITS-Nitazoxanide for Norovirus in Transplant Patients Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-0092
Record Dates: First submitted 2018-01-04; First posted 2018-01-10 (Actual); Results first posted 2022-10-24 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2021-06-25

CONDITIONS: Gastroenteritis Norovirus
Keywords: Efficacy; Hematopoietic Stem Cell; Nitazoxanide; Norovirus; Prospective, Randomized, Double-Blind Study; Safety; Solid Organ Transplant Recipients; Treatment
MeSH Terms: interventions — nitazoxanide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitazoxanide Arm (Experimental): 500 mg (one tablet) nitazoxanide by mouth twice daily with food for 56 consecutive doses. N=80
  Interventions: Drug: Nitazoxanide
- Placebo Arm (Placebo Comparator): Placebo (one tablet) by mouth twice daily with food for 56 consecutive doses. N=80
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nitazoxanide — One 500 mg tablet twice daily with food for 56 consecutive doses
  Arms: Nitazoxanide Arm
Other: Placebo — One tablet twice daily with food for 56 consecutive doses
  Arms: Placebo Arm

SUMMARY:
This is a phase 2 multi-center, double-blind, placebo-controlled study of the efficacy and safety of nitazoxanide for the treatment of solid organ and hematopoietic stem cell transplant recipients with symptomatic diarrhea due to Norovirus. The study involves a total of 160 Hematopoietic Stem Cell or Solid Organ transplant recipients, equal to or greater than 12 years of age with diagnosis of Norovirus who will be selected and randomly assigned (1:1) to nitazoxanide or placebo group. The study duration is 60 months and subject participation duration is 6 months. Given the safety of prolonged therapy with nitazoxanide, lack of interactions with common post-transplant medications, putative antiviral activity and prolonged duration of viral shedding we are assessing 56 doses of therapy. The longitudinal monitoring phase will provide useful information on the course of host and viral responses in subjects with chronic Norovirus infection with and without treatment. Randomization will be stratified by age group (pediatric (12 through 17 years) vs. adult (greater than or equal to 18 years)), chronicity of Norovirus-associated symptoms (acute (less than 14 days) vs. chronic (greater than or equal to 14 days)) and transplant type (solid organ (SOT)) vs. hematopoietic stem cell transplant (HSCT)). Enrolled subjects will participate in 2 phases of the study: Treatment Phase, which will include dosing with the assigned study agent for 28 days. Longitudinal Monitoring Phase which will include telephone call on Days 35, 53, 113, 173. Primary objective is 1) to assess the clinical efficacy of nitazoxanide for the management of acute and chronic Norovirus in transplant recipients.

DETAILED DESCRIPTION:
This is a phase 2 multi-center, double-blind, placebo-controlled study of the efficacy and safety of nitazoxanide for the treatment of solid organ and hematopoietic stem cell transplant recipients with symptomatic diarrhea due to Norovirus. The study involves a total of 160 Hematopoietic Stem Cell or Solid Organ transplant recipients, equal to or greater than 12 years of age with diagnosis of Norovirus who will be selected and randomly assigned (1:1) into two treatment groups: nitazoxanide or placebo. The study duration is approximately 60 months and subject participation duration is approximately 6 months. Given the safety of prolonged therapy with nitazoxanide, lack of interactions with common post-transplant medications, putative antiviral activity and prolonged duration of viral shedding we are assessing 56 doses of therapy. The longitudinal monitoring phase will provide useful information on the course of host and viral responses in subjects with chronic Norovirus infection with and without treatment. Randomization will be stratified by age group (pediatric (12 through 17 years) vs. adult (greater than or equal to 18 years)), chronicity of Norovirus-associated symptoms (acute (less than 14 days) vs. chronic (greater than or equal to 14 days)) and transplant type (solid organ (SOT)) vs. hematopoietic stem cell transplant (HSCT)). Enrolled subjects will participate in 2 phases of the study: Treatment Phase, which will include dosing with the assigned study agent for 28 days. Longitudinal Monitoring Phase which will include telephone call on Days 35, 53, 113, 173. Primary objective is 1) to assess the clinical efficacy of nitazoxanide for the management of acute and chronic Norovirus in transplant recipients. Secondary Objectives are 1) to assess the virologic efficacy of nitazoxanide and 2) to assess the safety of nitazoxanide for the management of acute and chronic Norovirus in transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

Subjects should meet all of the following inclusion criteria:

1. Male or female age > / = 12 years.
2. Recipient of a solid organ or hematopoietic stem cell transplant.
3. Positive test result for Norovirus within 14 days of enrollment that is obtained as part of routine clinical care using a Norovirus testing available to the site.
4. Active GI symptoms (diarrhea, or vomiting) that, in the opinion of the PI, are secondary to Norovirus. Patients must have active diarrhea, which is defined as at least 3 days of Bristol 6 or 7 stools in the past 2 weeks prior to enrollment per patient report.
5. Willing and able to provide written informed consent and assent before initiation of any study procedures, consistent with local IRB policy.
6. Subjects must be of non-childbearing potential or if of childbearing potential, must be using an effective method of birth control or must be abstinent.

   * Non-childbearing potential is defined as surgically sterile or postmenopausal for > one year.
   * Effective methods of birth control include the use of hormonal or barrier birth control such as implants, injectable contraceptives, combined oral contraceptives, intrauterine devices (IUDs),or condoms with spermicidal agents during study period. Female subjects must be using an effective method of birth control or practice abstinence and must agree to continue such precautions during the study and for 30 days after the Day 28 study visit.
   * A woman is eligible if she is monogamous with a vasectomized male.This subject is considered low risk and not required to use contraception.
7. Agrees to complete all screening requirements, study visits and procedures.

Exclusion Criteria:

Subjects meeting any of the exclusion criteria at baseline will be excluded from study participation:

1. Other identified infectious causes of diarrhea at screening. Alternative diagnosis requiring treatment would be considered a co-infection; if the testing is positive for a pathogen that the PI does not feel is causing the symptoms, they may be included but the PI or his/her designee must document that the positive test is not clinically significant, does not require treatment and is not causing the symptoms making the patient eligible for enrollment.
2. Any condition that would, in opinion of the Site Investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
3. Subjects receiving oral or intravenous immunoglobulin therapy concurrently or in the 14 days prior to enrollment.
4. Nitazoxanide use for any illness in the previous 30 days prior to randomization.
5. Have received experimental products within 30 days prior to the study entry or plan to receive experimental products at any time during the study
6. Known sensitivity to nitazoxanide or any of the excipients comprising the nitazoxanide tablets.
7. Subjects unable to swallow oral medications.
8. Subjects with ostomy.
9. Women who are pregnant or lactating or have a positive urine pregnancy test at screening/enrollment/Day 1.

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Northwestern University - Comprehensive Transplant Center, Chicago, Illinois
  - University of Kansas Medical Center - Infectious Diseases, Kansas City, Kansas
  - Johns Hopkins Hospital - Medicine - Infectious Diseases, Baltimore, Maryland
  - University of Michigan School of Public Health - Epidemiology, Ann Arbor, Michigan
  - University of Michigan - Infectious Disease Clinic at Taubman Center, Ann Arbor, Michigan
  - University of Nebraska Medical Center - Infectious Diseases, Omaha, Nebraska
  - Cincinnati Children's Hospital Medical Center Vaccine Research Center, Cincinnati, Ohio
  - University of Pittsburgh - Medicine - Infectious Diseases, Pittsburgh, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC - Pediatric Infectious Diseases, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center - Internal Medicine Subspecialties Clinic, Dallas, Texas
  - Fred Hutchinson Cancer Research Center - Vaccine and Infectious Diseases, Seattle, Washington
  - University of Washington - Medicine, Seattle, Washington

REFERENCES:
- [Derived] Shawar S, Concepcion BP. A Gut-Wrenching Infection: Norovirus in a Kidney Transplant Recipient. Clin J Am Soc Nephrol. 2023 Sep 1;18(9):1231-1233. doi: 10.2215/CJN.0000000000000243. Epub 2023 Jun 29. No abstract available. PMID 37382971

RESULTS

PARTICIPANT FLOW:
Groups:
- Nitazoxanide (500 mg): A single 500 mg tablet of nitazoxanide administered orally twice daily with food for 56 consecutive doses over 28 days.
  Nitazoxanide: a synthetic antiprotozoal agent, chemically designated as 2-acetyloxy-N-(5-nitro-2-thiazolyl) benzamide. Nitazoxanide will be supplied as 500 mg round, yellow, film-coated tablets.
- Placebo: A single matching placebo tablet administered orally twice daily with food for 56 consecutive doses over 28 days.
  Placebo: a round, yellow, film-coated tablet with the same inactive ingredients as the nitazoxanide tablet. The placebo tablet will be formulated for the same appearance as nitazoxanide.
Period: Overall Study
Arm/Group | Nitazoxanide (500 mg) | Placebo
Started | 16 | 15
Completed | 12 | 10
Not Completed | 4 | 5
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — COVID-19 Pandemic | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Nitazoxanide (500 mg): A single 500 mg tablet of nitazoxanide administered orally twice daily with food for 56 consecutive doses over 28 days.
- Placebo: A single matching placebo tablet administered orally twice daily with food for 56 consecutive doses over 28 days.
- Total: Total of all reporting groups
Arm/Group | Nitazoxanide (500 mg) | Placebo | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (10.7) | 55.8 (14.0) | 57.4 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 11 | 13 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Duration of symptoms [Count of Participants; unit: Participants] — Duration of symptoms in days. Acute duration is defined as fewer than 14 days. Chronic duration is defined as 14 or more days.
  Participants
    Acute | 4 | 3 | 7
    Chronic | 12 | 12 | 24
Transplant type [Count of Participants; unit: Participants]
  Solid organ | 15 | 15 | 30
  Hematopoietic Stem Cell Transplant | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Initial Clinical Resolution of Norovirus Symptoms
Description: Time (in days) from randomization until the study day when clinical resolution occurred. Clinical resolution was assessed from participant's daily diaries and was defined as cessation of vomiting and no stools classified by the Bristol Stool Chart as diarrhea (Type 6 or 7) for at least 48 hours.
Time Frame: 48 hours through Day 180
Population: Modified Intention-to-Treat (mITT) Population: The mITT population included all randomized participants who received at least one dose of assigned study drug. Analyses were performed according to randomized treatment assignment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Nitazoxanide (500 mg) | Placebo
Number analyzed (Participants) | 16 | 15
days | 19 [1 to 31] | 11 [2 to 14]
Statistical Analysis 1: Comparison: Nitazoxanide (500 mg) vs Placebo; The null hypothesis is that there is no difference in time until clinical resolution between study arms, with a two-sided alternative; Test type: Superiority; p = 0.459, Likelihood Ratio Test — No adjustment for multiple comparisons was made. The a priori threshold for statistical significant is 0.05; The null hypothesis is that there is no difference in time until clinical resolution between study arms, with a two-sided alternative; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.33 to 1.64] — HR estimated from a Cox model

2. Secondary Outcome: Number of Participants Experiencing Laboratory Adverse Events (AEs)
Description: Participants experiencing at least one new laboratory adverse event. Laboratory parameters include White Blood Cell (WBC), Hemoglobin, Platelet Count, Creatinine, Alkaline Phosphatase, Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Blood Urea Nitrogen (BUN), and Bilirubin. Laboratory results were considered AEs using the following thresholds : WBC greater than the upper limit of normal (ULN), hemoglobin less than the lower limit of normal (LLN), platelet count less than the LLN; creatinine greater than the ULN; alkaline phosphatase greater than the ULN; ALT greater than the ULN, AST greater than the ULN, BUN greater than or equal to the ULN, and bilirubin greater than the ULN. ULN and LLN values differed by site, sex, and age category.
Time Frame: Day 1 (baseline) through Day 60
Population: Safety Population: The safety population includes all participants who were randomized and received at least one dose of study treatment. Analyses are performed according to treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Nitazoxanide (500 mg) | Placebo
Number analyzed (Participants) | 16 | 15
Participants | 11 | 13

3. Secondary Outcome: Change in Viral Titer (Day 1 to Day 180)
Description: Change in viral titer defined as the difference between the Day 180 viral titer and the Day 1 viral titer. Participants were analyzed for the viral load test type (Norovirus GII or Norovirus GI) that they tested positive for at baseline (Day 1).
Time Frame: Day 1 (baseline) and Day 180
Population: Modified Intention-to-Treat (mITT) Population: The mITT population included all randomized participants who received at least one dose of assigned study drug. Only participants with results at Days 1 and 180 were included. No participants in Placebo GI subgroup had results at both days. Analyses were performed based on randomized treatment assignment. Fewer than 5 participants per treatment arm tested positive for Norovirus GI at baseline thus no GI specific statistical analyses were conducted.
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | Nitazoxanide (500 mg) | Placebo
Number analyzed (Participants) | 11 | 9
titer
  Norovirus GII: number analyzed (Participants) | 9 | 9
  Norovirus GII | -3.9 (9.8) | -4.2 (6.8)
  Norovirus GI: number analyzed (Participants) | 2 | 0
  Norovirus GI | -11.4 (3.5) |
Statistical Analysis 1: Comparison: Nitazoxanide (500 mg) vs Placebo; Includes participants in the Norovirus GII subgroup. The null hypothesis is that there is no difference in time until clinical resolution between study arms, with a two-sided alternative; Test type: Superiority; p = 0.735, ANCOVA — No adjustment for multiple comparisons was made. The a priori threshold for statistical significant is 0.05; Titer values were log-transformed

4. Secondary Outcome: Number of Participants Reporting Hospitalization
Description: Hospitalizations included any admission to a hospital for treatment and were not reported as Serious Adverse Events (SAEs).
Time Frame: Day 1 (baseline) through Day 60
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nitazoxanide (500 mg) | Placebo
Number analyzed (Participants) | 16 | 15
Participants | 4 | 7

5. Secondary Outcome: Number of Participants Reporting Protocol-Specified SAEs
Description: Protocol-specified SAEs included any adverse event or suspected adverse reaction which, in the view of the investigator or sponsor, resulted in any of the following: death, life threatening adverse event, persistent or significant disability or incapacity or substantial disruption of the ability to conduct normal life function, congenital anomaly or birth defect, or an important medical event that may jeopardize the participant and require medical or surgical intervention. Hospitalizations were collected as a secondary outcome measure and were not reported as SAEs.
Time Frame: Day 1 (baseline) through Day 60
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nitazoxanide (500 mg) | Placebo
Number analyzed (Participants) | 16 | 15
Participants | 0 | 2

6. Secondary Outcome: Number of Participants Experiencing Unsolicited Non-Serious Adverse Events
Description: Unsolicited adverse events were defined as any non-serious clinical adverse events that were not collected as clinical outcome measures and resulted in either modification in the administration of study drug or discontinuation of the study drug.
Time Frame: Day 1 (baseline) through Day 60
Population: Unsolicited adverse events were defined as any non-serious clinical adverse events that were not collected as clinical outcome measures and resulted in either modification in the administration of study drug or discontinuation of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Nitazoxanide (500 mg) | Placebo
Number analyzed (Participants) | 16 | 15
Participants | 2 | 0

7. Secondary Outcome: Time to First Negative Viral Load
Description: Time (in days) from randomization until the first study day the participant had either a negative result or a result less than the lower limit of quantitation (LLOQ) for the viral load test type (Norovirus GII or Norovirus GI) that they initially tested positive for at baseline. Participants were analyzed for the viral load test type (Norovirus GII or Norovirus GI) that they tested positive for at baseline (Day 1).
Time Frame: Day 1 (baseline) and Day 180
Population: Modified Intention-to-Treat (mITT) Population: The mITT population included all randomized participants who received at least one dose of assigned study drug. Only participants who tested positive at Day 1 were included. Analyses were performed based on randomized treatment assignment. Fewer than 5 participants per treatment arm tested positive for Norovirus GI at baseline thus no GI specific statistical analyses were conducted.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Nitazoxanide (500 mg) | Placebo
Number analyzed (Participants) | 14 | 15
days
  Norovirus GII: number analyzed (Participants) | 12 | 12
  Norovirus GII | NA [45 to NA] — Estimates were not calculable due to an insufficient number of participants (less than 50% of participants/treatment group) having a negative viral load. | NA [120 to NA] — Estimates were not calculable due to an insufficient number of participants (less than 50% of participants/treatment group) having a negative viral load.
  Norovirus GI: number analyzed (Participants) | 2 | 3
  Norovirus GI | NA [12 to NA] — Estimates were not calculable due to an insufficient number of participants (less than 50% of participants/treatment group) having a negative viral load. | 22 [13 to NA] — Estimates were not calculable due to an insufficient number of participants (less than 50% of participants/treatment group) having a negative viral load.
Statistical Analysis 1: Comparison: Nitazoxanide (500 mg) vs Placebo; Includes participants in the Norovirus GII subgroup. The null hypothesis is that there is no difference in time until first negative viral load between study arms, with a two-sided alternative; Test type: Superiority; p = 0.873, Likelihood Ratio Test — No adjustment for multiple comparisons was made. The a priori threshold for statistical significance is 0.05; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.19 to 4.06]

ADVERSE EVENTS:
Time Frame: 180 days
Arm/Group | Nitazoxanide (500 mg) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 2/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 2/15
Other Adverse Events (participants affected / at risk) | 12/16 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitazoxanide (500 mg) (N=16) | Placebo (N=15)
Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Uremia (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitazoxanide (500 mg) (N=16) | Placebo (N=15)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 2 (2) | 1 (2)
Aspartate Aminotransferase Increased (Investigations) | 2 (2) | 3 (4)
Blood Alkaline Phosphatase Increased (Investigations) | 2 (4) | 3 (6)
Blood Bilirubin Increased (Investigations) | 1 (1) | 2 (4)
Blood Creatinine Increased (Investigations) | 6 (10) | 3 (3)
Blood Urea Increased (Investigations) | 7 (13) | 3 (6)
Haemoglobin Decreased (Investigations) | 3 (3) | 5 (6)
Platelet Count Decreased (Investigations) | 3 (3) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 1 (1) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
White Blood Cell Count Increased (Investigations) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT03395405/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT03395405/SAP_001.pdf